CLINICAL TRIAL: NCT05272319
Title: Genetic Collection Protocol
Status: Recruiting | Type: Observational
Sponsor: Arbor Research Collaborative for Health (Other)
Responsible Party: Sponsor
Other Study IDs: Genetic Collection - ChiLDReN
Record Dates: First submitted 2021-12-13; First posted 2022-03-09 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Liver Diseases
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Participants will have one-time collection of whole blood or saliva for DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study involves the one-time collection of whole blood or saliva samples for the extraction and storage of DNA for use in ongoing and future ChiLDReN studies.

DETAILED DESCRIPTION:
The purpose of this study is to establish a mechanism to collect a genetic biosample from the participants previously enrolled into clinical research under ChiLDReN-supported protocols (PROBE and BASIC). The samples will be linked to the data previously collected on the participant. Samples will be stored in the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) specimen repository and will be used in ongoing and future Network and Ancillary Studies of ChiLDReN to further address the pathophysiology and outcomes of these liver diseases.

ELIGIBILITY:
Inclusion Criteria:

* For Child Participants

  1. Previous enrollment in PROBE or BASIC
  2. Exited from one of the aforementioned studies.
  3. Consent for DNA sample collection obtained during enrollment during enrollment to one of the aforementioned studies but sample not previously collected.
  4. Still followed at the clinical site.

     Exclusion Criteria:

  <!-- -->

  1. Participant is deceased
  2. Participant exited from prior study due to violating eligibility criteria
  3. Participant cannot be contacted

Ages: 24 Hours to 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: The eligible study population are those child participants who signed consent to participate in a prior research study that collects DNA biospecimens and for whom the specimen was never obtained. If those participants are still followed by the site.
Sampling Method: Probability Sample
Enrollment: 2230 (Estimated)
Dates: Start 2022-04-06 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Augment a repository of DNA | beginning of study through study completion, an average of 1 year.
  The major objective of this protocol is to augment a repository of DNA from participants previously enrolled into clinical research but for whom a DNA biosample was not previously collected. The acquisition and storage of DNA from participants will make available an important resource for future and ongoing studies that may evaluate etiology, pathogenesis, biomarkers, pharmacogenomics, and genetic modifiers of these rare disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Ed Doo, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK); Katrina Loh, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK); John Magee, MD, Principal Investigator — University of Michigan; Lisa Henn, PhD, Principal Investigator — Arbor Research Collaborative for Health
Locations (13):
- United States (12):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Lurie Children's Hospital, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Texas Children's Hospital; Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No